CLINICAL TRIAL: NCT00587704
Title: Paravertebral Blocks Techniques: A Pilot Study to Compare Nerve Stimulation vs. Anatomic Landmarks for Patients Undergoing Inguinal Hernia Repair
Brief Title: Paravertebral Blocks: Pilot Study to Compare Nerve Stimulation vs. Anatomic Landmarks in Inguinal Hernia Repair
Acronym: PVB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Steven R. Clendenen, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 07-002759
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Nerve Stimulation (Other): Use of nerve stimulator for placement of PVB nerve block
  Interventions: Procedure: PVB using nerve stimulation
- Anatomic landmarks (Other): Use of anatomic landmarks for placement of PVB block
  Interventions: Procedure: PVB using anatomic landmarks

INTERVENTIONS:
Procedure: PVB using nerve stimulation — 5ml of 1% ropivacaine injected incrementally
  Arms: Nerve Stimulation
Procedure: PVB using anatomic landmarks — 5ml of 1% ropivacaine injected incrementally
  Arms: Anatomic landmarks

SUMMARY:
Primary aim:

1. To compare the nerve stimulation vs. anatomic techniques of paravertebral block of T11-L1 in providing surgical anesthesia for patients undergoing inguinal hernia repair.

Secondary aims:

1. Compare VAS pain scores in the two groups of patients over the first 24 hours.
2. Compare opioid intake over the first 24 hours in the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral open inguinal herniorrhaphy
* Patient must be >18 years of age
* ASA physical status of I, II, or III
* Patient competent to provide informed consent

Exclusion Criteria:

* Patient < 18 years of age
* Pregnant or lactating women
* Patient unwilling or unable to provide informed consent
* Contraindications to regional anesthesia
* Allergy to amide local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Successful full block at T11-L1 | Every 10 minutes until full block achieved

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Clendenen, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States